CLINICAL TRIAL: NCT06711302
Title: Remote Ischemic Conditioning for Efficacy in Patients With Aneurysmal Subarachnoid Hemorrhage: a Multi-center, Randomized, Double-blind, Sham-controlled, Parallel-group Trial
Brief Title: Remote Ischemic Conditioning for Efficacy in Patients With Aneurysmal Subarachnoid Hemorrhage
Acronym: REPAIR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HX-A-2024009
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Subarachnoid Hemorrhage; Cerebrovascular Disorders; Brain Diseases; Stroke; Cardiovascular Diseases; Vascular Diseases; Nervous System Diseases
MeSH Terms: conditions — Subarachnoid Hemorrhage; Cerebrovascular Disorders; Brain Diseases; Stroke; Cardiovascular Diseases; Vascular Diseases; Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham group (Sham Comparator): Guideline-based therapy+Sham RIC is given twice a day with 60mmHg pressure.
  Interventions: Device: Sham RIC
- RIC Group (Experimental): Guideline-based therapy+RIC RIC is given twice a day with 200mmHg pressure.
  Interventions: Device: Remote Ischemic Conditioning treatment instrument

INTERVENTIONS:
Device: Sham RIC — Remote Ischemic Conditioning is given twice a day with 60mmHg pressure.
  Arms: Sham group
Device: Remote Ischemic Conditioning treatment instrument — Remote Ischemic Conditioning is given twice a day with 200mmHg pressure.
  Arms: RIC Group

SUMMARY:
Several recent large-scale clinical trials aimed at improving subarachnoid hemorrhage(SAH) outcomes have concluded with negative results, failing to enhance the prognosis for these patients. Consequently, there is an urgent demand for novel treatment strategies and approaches to address the challenges posed by SAH.

Remote ischemic conditioning(RIC) has gained considerable attention in the treatment of stroke, particularly ischemic stroke, with numerous studies demonstrating its potential to enhance neurological outcomes compared to conventional treatments alone.RIC for the treatment of SAH is an investigative strategy in its initial stages. The neuroprotective effects of RIC, particularly its potential to preserve cranial nerve function and ameliorate neurological deficits, confer significant value in the treatment of SAH patients.

The precise manner in which SAH patients may benefit from RIC treatment, and the mechanisms by which it improves neurological function, remain to be fully understood. Consequently, randomized controlled trials are necessary to validate the efficacy of RIC in this patient population and to delineate the optimal therapeutic protocols for its application.

Based on the above discussion, this study aims to explore the efficacy and safety of RIC in the treatment of SAH.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with aneurysmal subarachnoid hemorrhage confirmed by imaging examination (diagnosed by computed tomography and confirmation of an intracranial aneurysm by CT angiography or digital subtraction angiography);
2. The Hunt-Hess grade is 2-3 at admission;
3. Onset of aneurysmal subarachnoid hemorrhage ≤72 hours;
4. The responsible aneurysm has been treated by endovascular interventional therapy;
5. 18≤ age ≤80 years old;
6. Informed consent must be obtained from participants or legally authorized representatives.

Exclusion Criteria:

1. Patients with other intracerebral hemorrhage or other types of subarachnoid hemorrhage;
2. Previous neurological deficits (mRS Score ≥1) or psychiatric disorders that can confound neurological or functional assessments;
3. With severe comorbidities and a life expectancy of less than 90 days;
4. Refractory hypertension (Systolic blood pressure> 180 mmHg or diastolic blood pressure >110 mmHg);
5. Contraindications of RIC: severe soft tissue injury of the lower limbs, etc;
6. Concurrent participation in another protocol investigating a different experimental therapy;
7. Any condition that the investigator believes may increase the patient's risk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of mRS (0-2) | 90±7 days
  Modified Rankin Scale, mRS; min:0, max:6; A smaller score indicates a better prognosis.

SECONDARY OUTCOMES:
Proportion of mRS (0-1) | 90±7 days
  Modified Rankin Scale, mRS; min:0, max:6; A smaller score indicates a better prognosis.
mRS Score as ordinal variable | 7±1 days
  Modified Rankin Scale, mRS; min:0, max:6; A smaller score indicates a better prognosis.
mRS Score as ordinal variable | 30±7 days
  Modified Rankin Scale, mRS; min:0, max:6; A smaller score indicates a better prognosis.
Cognitive function score as ordinal variable | 7±1 days
  Montreal Cognitive Assessment, MoCA. The total score is 30, with higher scores indicating better cognitive function.
The complete blood count | During hospitalization
  up to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data and study materials will be accessible.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the main trial results, subject to legal and ethical approvals.
Access Criteria: Approved investigators will have access to deidentified data by contacting the corresponding author.

REFERENCES:
- [Derived] Jin T, Niu H, Liu L, Yin Y, Zhao W, Feng X, Xu L, Hess DC, Liu A, Ji X. Remote ischaemic conditioning for efficacy in patients with aneurysmal subarachnoid haemorrhage (REPAIR): protocol for a multicentre, randomised, double-blind, sham-controlled, parallel-group trial. BMJ Open. 2025 Aug 11;15(8):e101350. doi: 10.1136/bmjopen-2025-101350. PMID 40789732